CLINICAL TRIAL: NCT00908921
Title: Efficacy and Safety of Glimepiride as Oral Anti-Diabetic (OAD) Initiation Mono- Therapy in Chinese Type 2 Diabetes Mellitus (T2DM)
Brief Title: Efficacy and Safety of Glimepiride as Oral Anti-Diabetic (OAD) Initiation Mono-therapy in Chinese Type 2 Diabetes Mellitus (T2DM)
Acronym: GREAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLIME_L_04409
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride

ARMS (1):
- 1 (Experimental): The treatment period is 16 weeks with 5 visits: at weeks 2, 4, 8, 12, 16. At every visit if Fasting Blood Glucose (FBG) >7.0mmol/L the Glimepiride dosage is increased from 1mg to 2mg or 2mg to 4mg.
  At every visit if FBG<3.9mmol/L the Glimepiride dosage is decreased from 4mg to 2mg or 2mg to 1mg.
  Patients who have been on 4mg for 4 weeks and FBG>11.0mmol/L at visit, another treatment can be added at the physician's discretion.
  Interventions: Drug: GLIMEPIRIDE

INTERVENTIONS:
Drug: GLIMEPIRIDE — Dosage of 1mg, 2mg and 4mg of AMARYL (Glimepiride)

SUMMARY:
To investigate the glycosylated hemoglobin (HbA1c) control of Glimepiride (AMARYL) as OAD initiation mono-therapy in type 2 diabetic patients in China.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed T2DM and inadequately controlled with diet and exercise or T2DM diagnosed <6 months and who had not taken oral antidiabetic medication or insulin for >3months.
* HbA1C more than 7.5 and less than 11.

Exclusion Criteria:

* Fasting plasma glucose of >13.5mmol/L
* Type 1 Diabetes Mellitus (T1DM)
* Patient with acute illness hospitalized in last 2 months
* Patient with active liver disease, impaired renal or hepatic functions
* Known hypersensitivity to glimepiride, other sulfonylureas, other sulfonamides or any other excipients of AMARYL
* Pregnant and lactating women

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2009-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change in glycosylated hemoglobin (HbA1c) rate | week 16

SECONDARY OUTCOMES:
Fasting Plasma Glucose (FPG) rate | week 16
Post Prandial Glucose (PPG) rate | week 16
Percentage of patients achieving HbA1c <7.0 | week 16

CONTACTS AND LOCATIONS:
Overall Officials: Mei Mao, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Shanghai, China

REFERENCES:
- [Derived] Guo XH, Lv XF, Han P, Zhang XZ, Yang HZ, Duan WR, Gao Y. Efficacy and safety of glimepiride as initial treatment in Chinese patients with Type 2 diabetes mellitus. Curr Med Res Opin. 2013 Mar;29(3):169-74. doi: 10.1185/03007995.2013.765396. Epub 2013 Jan 24. PMID 23305037